CLINICAL TRIAL: NCT04096729
Title: Patients Commitment to Compression Therapy
Acronym: POMP
Status: Completed | Type: Observational
Sponsor: Belarusian State Medical University (Other)
Responsible Party: Principal Investigator, Ihar Ihnatovich, Professor, Belarusian State Medical University
Other Study IDs: 1-30082019
Record Dates: First submitted 2019-09-16; First posted 2019-09-20 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Compression; Vein; Patient Satisfaction
Keywords: commitment to treatment; compression stockings; varicose veins
MeSH Terms: conditions — Patient Satisfaction; Varicose Veins | interventions — Stockings, Compression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients who have consulted and need compression therapy using: 1) age from 18 to 75 years; 2) compression therapy prescribed by a phlebologist. The exclusion criterion is hearing impairment, which could interfere with a telephone questionnaires.
  Interventions: Other: compression stockings

INTERVENTIONS:
Other: compression stockings — patients will be prescribed compression therapy for varicose veins of the legs using compression stockings

SUMMARY:
The study Patients Commitment to compression therapy (POMP) is observational, prospective. After the Phlebologist consultation after 1 month and 1 year, a telephone questionnaire is carried out for the patients included in the study with the involvement of a company specializing in conducting a telephone questionnaire. Patients will be interviewed about the implementation of the doctor's recommendations regarding compression therapy over a period 1 month and 1 year.

DETAILED DESCRIPTION:
Phlebologists will include in the study patients who have consulted and need compression therapy using a compression hosiery. Patients are recommended compression hosiery that meet RAL-GZ 387, Oeko-Tex Standart 100. At the same time, the design of this study does not provide for restrictions on the acquisition by patients of other type compression hosiery.

Inclusion of patients in the study is carried out only after obtaining written informed consent from them for data registration and subsequent telephone questionnaires. Demographic, anamnestic, sociological data, such as educational level, labor characteristics (heavy physical labor, prolonged orthostasis, prolonged sitting position) recorde in the patient's individual card. Women provide information on the number of births, menopause, use of hormone replacement therapy at the time of the study. A diagnosis performed for each lower limb according to only the clinical part of the CEAP classification without other details. The phlebologist individually for each patient determines the mode of wearing compression hosiery. In addition to compression therapy, it is possible to prescribe any other type of drug and / or surgical treatment. In the subsequent analysis, data on the lower limb with more severe manifestations of venous insufficiency are used.

Table 1. Main characteristics of the patients included in the study Class С Age, years Sex Мail/Femail University education Yes / No Prolonged orthostasis Yes / No Hard physical labor Yes / No Prolonged sitting position Yes / No Family history of Chronic Vein Disease Yes / No A history of Venous Thromboembolism Yes / No Smoking Yes / No History of childbirth (among women) Number 0-…. Hormonal contraception / hormone replacement therapy (among women) Yes / No

1 month and 1 year after the consultation patients will interrogate about the implementation of the doctor's recommendations regarding compression therapy (Tabl. 2) Table 2. Questions included in the telephone survey You have been prescribed compression hosiery. Have you bought it?

* Did not buy
* Bought immediately after a visit to the doctor
* Not immediately bought (after how many days) Which product did you buy?
* Knee socks
* Stockings
* One-leg stocking with zipper at the waist (monostocking)
* Tights Do you follow the recommended doctor's regimen for wearing compression hosiery? - ---
* Yes
* No

If you did not comply with the compression hosiery pattern, then why?

* Too difficult to put on / take off
* Uncomfortable to wear
* Hot to wear
* Itching when used
* Ugly
* Does not help
* It gets worse when I start wearing
* I can not wash the product every day
* Other (with explanation) Did you wear compression hosiery before being included in the study?
* Yes
* No What kind of compression hosiery had you wear before you entered the study?
* Knee socks
* Stockings
* One-leg stocking with zipper at the waist (monostocking)
* Tights Compression class
* 1
* 2
* 3

How are you satisfied with the effect of the using compression hosiery? Score in points from 0 to 10, where 10 is the maximum level of satisfaction

How are you satisfied with the comfort of the using compression hosiery? Score in points from 0 to 10, where 10 is the maximum level of satisfaction

How are you satisfied with the quality of the using compression hosiery? Score in points from 0 to 10, where 10 is the maximum level of satisfaction

ELIGIBILITY:
Inclusion Criteria:

* varicose veins of the legs and compression therapy prescribed by a phlebologist

Exclusion Criteria:

* hearing impairment, which could interfere with a telephone questionnaires

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with varicose veins of the legs
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-01-26 (Actual)

PRIMARY OUTCOMES:
number of patients who will follow prescribed compression therapy and recommended doctor's regimen for wearing compression hosiery | 1 month
  1-followed 2- did not followed
number of patients who will follow prescribed compression therapy and recommended doctor's regimen for wearing compression hosiery | 1 year
  1-followed 2- did not followed

SECONDARY OUTCOMES:
number of patients who will satisfy with the effect,comfort and quality of the using compression hosiery | 1 month
  Score in points from 0 to 10, where 10 is the maximum level of satisfaction
number of patients who will satisfy with the effect,comfort and quality of the using compression hosiery | 1 year
  Score in points from 0 to 10, where 10 is the maximum level of satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Ihar Ihnatovich, Prof, Principal Investigator — Belarusian State Medical University
Locations (2):
- Belarus (2):
  - Educational Institution"Belarusian State Medical University", Minsk, Dzerzhinski Ave., 83
  - Belarusian State Medical University, Minsk

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wittens C, Davies AH, Baekgaard N, Broholm R, Cavezzi A, Chastanet S, de Wolf M, Eggen C, Giannoukas A, Gohel M, Kakkos S, Lawson J, Noppeney T, Onida S, Pittaluga P, Thomis S, Toonder I, Vuylsteke M, Esvs Guidelines Committee, Kolh P, de Borst GJ, Chakfe N, Debus S, Hinchliffe R, Koncar I, Lindholt J, de Ceniga MV, Vermassen F, Verzini F, Document Reviewers, De Maeseneer MG, Blomgren L, Hartung O, Kalodiki E, Korten E, Lugli M, Naylor R, Nicolini P, Rosales A. Editor's Choice - Management of Chronic Venous Disease: Clinical Practice Guidelines of the European Society for Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg. 2015 Jun;49(6):678-737. doi: 10.1016/j.ejvs.2015.02.007. Epub 2015 Apr 25. No abstract available. PMID 25920631
- [Background] Mosti G, Partsch H. Bandages or double stockings for the initial therapy of venous oedema? A randomized, controlled pilot study. Eur J Vasc Endovasc Surg. 2013 Jul;46(1):142-8. doi: 10.1016/j.ejvs.2013.04.015. Epub 2013 May 15. PMID 23683393
- [Background] Amsler F, Blattler W. Compression therapy for occupational leg symptoms and chronic venous disorders - a meta-analysis of randomised controlled trials. Eur J Vasc Endovasc Surg. 2008 Mar;35(3):366-72. doi: 10.1016/j.ejvs.2007.09.021. Epub 2007 Dec 11. PMID 18063393